CLINICAL TRIAL: NCT01384929
Title: Indian Intensive Care Case Mix and Practice Patterns Study
Brief Title: Study of Intensive Care Units in India
Acronym: INDICAPS
Status: Completed | Type: Observational
Sponsor: Indian Society of Critical Care Medicine (Other)
Responsible Party: JV Divatia / Chairman, Clinical Research, Dr. Rajesh Chawla, President, Indian Society of Critical Care Medicine
Other Study IDs: ISCCM01
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-04

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: All patients present in the ICU on the selected days

SUMMARY:
There is scant data on the casemix and practices in Indian intensive care units (ICUs). Most of the available data comes from single centre studies. There is a dire need to have data from Indian ICUs to reflect the vast spectrum of critical care illness, services and practices. INDICAPS planned to collect data of all patients in the ICU on one particular day, and four such days spread throughout a one-year period were selected: the second Wednesday of July and October this year, i.e. July 14 and October 13, 2010 and the second Wednesday of January and April next year, i.e. January 12 and April 13, 2011. As many ICUs all over the country as possible were asked to participate. The investigators aimed to gather information about ICUs, patients in ICUs, the types and severity of illness, monitoring and therapeutic modalities used, types of infections,mortality rates, etc.

DETAILED DESCRIPTION:
The following information will be analysed:

Case-mix, severity of illness, prevalence of infection, hemodynamic monitoring and therapy, mechanical ventilation practices, nutrition and outcome

* Seasonal and regional variations in the above
* Epidemiology and variations in antibiotic use
* Patterns of microorganisms and outcome
* Prevalence and outcome of specific tropical febrile illnesses, including malaria, dengue fever, leptospirosis, scrub typhus
* Prevalence and outcome of toxins and poisonings
* Relation of ICU and hospital organizational issues to prevalence of infection and outcome
* Organisation of intensive care services
* End of life - Ethical decisions

ELIGIBILITY:
Inclusion Criteria:

* All patients present in the ICU July 14, 2010, October 13, 2010, January 12, 2011 and April 13, 2011

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients present in the ICU July 14, 2010, October 13, 2010, January 12, 2011 and April 13, 2011
Sampling Method: Non-Probability Sample
Enrollment: 4236 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30-days

SECONDARY OUTCOMES:
ICU Length of stay | 30 days
  Stay in ICU till 30 days
Hospital length of stay | 30 days
  Stay in hospital till 30 days
Hospital survival | 30 days
  Survival at hospital discharge or at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jigeeshu Divatia, MD, Study Chair — Indian Society of Critical Care Medicine
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India